CLINICAL TRIAL: NCT02957916
Title: Vanderbilt Childhood Obesity Registry
Acronym: VCOR
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, MD, MSCI, Vanderbilt University Medical Center
Other Study IDs: 121345
Record Dates: First submitted 2016-10-31; First posted 2016-11-08 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Childhood Onset Obesity; Pediatric Obesity; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA sample collected once in the form of either saliva or 5 mL of blood
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to better understand early onset obesity and to identify patients in interested in future research studies, including clinical trials, we aim to develop a registry for patients with early onset obesity.

DETAILED DESCRIPTION:
Obesity is an epidemic effecting the pediatric population. Currently, 17% of children are classified as obese and 32% as overweight. Many of these children develop complications including type 2 diabetes, dyslipidemia, hypertension and hepatic steatosis. Obesity is a global epidemic that lacks effective treatment options. Obesity has many underlying causes including genetic predisposition and environmental factors. Understanding the genetic basis of obesity may allow for more precisely targeted interventions including specific dietary plans and pharmacologic treatments. The most common cause of genetic obesity is haploinsufficiency of the melanocortin-4 receptor (MC4R). In obese adult cohorts, the prevalence of pathogenic MC4R mutations is 1-2%. Commercial testing is available for many obesity syndromes, but the cost is high and charges are not always covered by insurance. Clinicians have little motivation to test patients for MC4R mutations as no treatments are available and it is not clear if genetic testing results change patient behavior. This particular lab and other groups are working to develop novel pharmacologic treatments for obesity syndromes, such as MC4R deficiency. In order to better understand early onset obesity and to identify patients in interested in future research studies, including clinical trials, the investigators aim to develop a registry for patients with early onset obesity.

ELIGIBILITY:
Inclusion Criteria:

1. BMI >97th percentile for age and gender before 6 years old
2. Able to give written, informed consent/assent

Exclusion Criteria:

1. Diagnosis of Prader-Willi syndrome
2. Use of exogenous steroids or other medications known to cause abnormal weight gain
3. Cushing's syndrome, untreated growth hormone deficiency or untreated hypothyroidism as an etiology for the obesity
4. Hypothalamic obesity (obesity due to a brain tumor, head trauma or other brain lesion)
5. Currently pregnant

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with a history of excessive weight gain.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-11; Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of genetic mutations in DNA analysis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with collaborators and on a case by case basis. Please contact Dr. Shoemaker for information.